CLINICAL TRIAL: NCT03723733
Title: Compensatory Brain Mechanisms for Amygdala-associated Cognitive Dysfunction: Potential Role of the Cortical Mirror Neuron System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Other Study IDs: UESTC-neuSCAN-28
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: amygdala; mirror neuron system; brain network

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Behavioral: screen high and low triat subjects — use a range of questionniares to screen screen high and low triat subjects (eg. Autism, Anxiety, Depression traits and social network size)

SUMMARY:
Identify if the mirror neuron system, or other networks, can compensate for amygdala dysfunction, using behavior and structural/functional MRI.

DETAILED DESCRIPTION:
In the present study, investigators aim to investigate amygdala dysfunction & potential compensation in individuals with high and low traits (e.g. Autism, Anxiety, Depression traits, Alexithymia), high and low stress or protective factors in the environment (social network, early life stress) and different molecular genetic make-up. On the neural level, functional and structural connectivity as well as task-related BOLD activation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* history of head injury
* claustrophobia;
* medical or psychiatric illness
* female subjects were pregnant or taking oral contraceptives.
* taking any form of medication and drunk any caffeine-containing beverages on the day of the experiment.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: sutduents from University of Electronic Science and Technology of China
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
brain activity and connectivity during social and cognitive tasks | 2 hours
  brain activity and connectivity was measured by the fMRI scanner

CONTACTS AND LOCATIONS:
Locations (1):
- China, Sichuan, Chengdu, Sichuan, China